CLINICAL TRIAL: NCT06773208
Title: A Phase 2 Study of Azacitidine and Venetoclax to Treat Acute Myeloid Leukemia Patients With Measurable Residual Disease Before an Allogeneic Stem Cell Transplant
Brief Title: A Study of Azacitidine and Venetoclax in People With Acute Myeloid Leukemia (AML)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24-347
Record Dates: First submitted 2025-01-08; First posted 2025-01-14 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Acute Myeloid Leukemia (AML)
Keywords: Azacitidine; Venetoclax; Allogeneic Stem Cell Transplant; 24-347
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Azacitidine; venetoclax

STUDY DESIGN:
Intervention Model Description: This is a single-arm, single center, phase II study.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Azacitidine and Venetoclax (Experimental): Cycle length: 28 days Azacitidine 75 mg/m2 daily, on days 1-7, given IV or SC (generally given IV in our institution) Venetoclax 400 mg orally daily on days 1-28
  Interventions: Drug: Azacitidine (AZC); Drug: Venetoclax

INTERVENTIONS:
Drug: Azacitidine (AZC) — 75 mg/m2 daily, on days 1-7, given IV or SC
Drug: Venetoclax — Venetoclax 400 mg orally daily on days 1-28

SUMMARY:
The purpose of this study is to find out if azacitidine and venetoclax are an effective treatment approach to get rid of or lower measurable residual disease (MRD) in people with acute myeloid leukemia (AML) who have received standard chemotherapy and are planning to have an allogeneic hematopoietic stem cell transplant (HSCT). Allogeneic HSCT, sometimes called a bone marrow transplant, involves receiving healthy blood-forming cells (stem cells) from a donor in order to replace the patient's immune system and lower the chances of the disease returning (relapse).

ELIGIBILITY:
Inclusion Criteria:

* 1. Adult patient ≥18 years of age at the time of signing the informed consent form (ICF). Legal Authorized Representatives (LAR) are permitted.

  2. Patient is willing and able to adhere to the study visit schedule and other protocol requirements.

  3. Patient has a confirmed diagnosis of de-novo AML (non-APL) as per World Health Organization (2022) guidelines. All (non-APL) subtypes of AML are permitted, irrespective of ELN risk category or mutational status.

  4. Patient has received 1-3 cycles of intensive chemotherapy for remission induction.

  5. Patient is in a morphologic remission, defined as less than 5% percent blasts seen by aspirate differential (or immunohistochemistry if no aspirate available) from bone marrow biopsy.

  6. Patient and is either in CR, or CR with partial count recovery, either CRi/CRh\^1.

  1CR= BM with <5% blasts, absence of circulating blasts; absence of extramedullary disease, absolute neutrophil count (ANC) ≥ 1000 cells/µL and platelet (PLT) count ≥ 100,000/µL. CRh = CR with ANC 500-1000 cells/µL and PLT 50,000-100,000 /µL. CRi = CR without meeting CRh criteria (residual neutropenia or thrombocytopenia).

  7. Patient has positive measurable residual disease (MRD) at or above a level of 0.1%, by flow cytometry (MFC) or in molecular cases (NPM1 mutated or one of the CBF translocations) RT-qPCR at or above 0.01%, as described above (see section 3.6). If RT-qPCR is not available, MFC will be allowed for determining eligibility for molecular patients (at or above 0.1%).

  8. Patient is eligible for intensive chemotherapy and immediate allogeneic transplant, with intention to proceed to transplant after trial intervention.

  9. Patient has an ECOG performance status of ≤3 10. Patient has adequate organ function defined as:
  1. Serum aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 x ULN
  2. Serum total bilirubin < 1.5 x ULN (or direct bilirubin normal in subjects with total bilirubin > 1.5 ULN). Except in cases of Gilbert's disease.
  3. Creatinine clearance greater than 30 mL/min based on the Cockroft-Gault glomerular filtration rate (GFR) estimation.

     11. Absence of active uncontrolled infection, heart failure or severe psychiatric or neurological disease.

     12. Females of childbearing potential may participate provided they have a negative serum pregnancy test at screening and a negative serum OR urine pregnancy test within two weeks of starting on treatment.

     13. Females of reproductive potential should use effective contraception during the study, and for 6 months after last dose of azacitidine. Males with female partners of reproductive potential should use effective contraception during treatment and for 3 months after.

     Exclusion Criteria:

     1. Patients with acute promyelocytic leukemia (APL) or relapsed/refractory AML 2. Blast crisis of chronic myeloid leukemia 3. Patient with 5% blasts or more by bone marrow aspirate differential (or IHC if no aspirate available) 4. Patient has received previous therapy with a venetoclax containing regimen. 5. Patient has presence of any other condition that may increase the risk associated with study participation, and in the opinion of the investigator, would make the patient inappropriate for entry into the study.

     6. Patient has active uncontrolled systemic fungal, bacterial, or viral infection.

     7. Patient had recent, significant venous or arterial thrombotic event that would necessitate full anticoagulation or dual anti-platelet therapy, including PE within 30 days prior to start of treatment or insertion of drug eluting stent within 6 months prior to start of treatment. Chronic indications for anticoagulation such as atrial fibrillation, can be included if CHADS2 score below 4.

     8. Patient has mechanical heart valve. 9. Patient had recent significant hemorrhagic episode, at the discretion of investigator.

     10. Patient has significant active cardiac disease within 6 months prior to start of study treatment.

     11. Patient is known to have dysphagia, short-gut syndrome, gastroparesis, or other conditions that limit the ingestion or gastrointestinal absorption of drugs administered orally.

     12. Female subject who is pregnant or lactating.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-01-07 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
rate of MRD conversion | 1 year
  MRD status will be assessed from end-of-cycle bone marrow aspirate, in all patients. MRD will be assessed by flow cytometry (MFC) or by RT-qPCR in molecular patients. This is a dichotomous variable of positive versus negative MRD, with a pre-defined threshold as described above, of 0.1% for MFC or 0.01% in molecular patients .

SECONDARY OUTCOMES:
degree of MRD decrease | 1 year
  will be summarized as median and interquartile range.

CONTACTS AND LOCATIONS:
Overall Officials: Eytan Stein, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering at Basking Ridge (All Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (All Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (All Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Suffolk-Commack (All Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (Limited Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York
  - Memorial Sloan Kettering Nassau (All Protocol Activities), Rockville Centre, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm